CLINICAL TRIAL: NCT00696410
Title: Pilot Study to Assess the Impact of Zinc Supplementation on Left Ventricular Remodeling, Function, and Oxidative Stress in Nonischemic Cardiomyopathy
Brief Title: The Impact of Zinc Supplementation on Left Ventricular Function in Nonischemic Cardiomyopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jennifer Cowger , MD, MS, Assistant Professor, study Coinvestigator, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM0001911; NIHT32-HL007853
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Heart Failure; Cardiomyopathies
Keywords: Heart Failure; Cardiomyopathy; Remodeling; Antioxidant; Zinc; Copper
MeSH Terms: conditions — Heart Failure; Cardiomyopathies | interventions — Zinc Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHF patients Given Zinc Acetate (Experimental): Patients with CHF received zinc acetate 50 mg po TID. This is a pre-post study
  Interventions: Drug: Zinc Acetate
- Healthy controls (No Intervention): Health controls; no zinc acetate administered.

INTERVENTIONS:
Drug: Zinc Acetate — Zinc acetate 50 mg po TID for 10 months. Dose will be titrated to achieve ceruloplasmin levels ~10-12.
  Other Names: Galzin (zinc acetata, Teva Pharmaceuticals)
  Arms: CHF patients Given Zinc Acetate

SUMMARY:
Heart failure affects over 5.3 million Americans and, while other cardiovascular diseases have enjoyed a reduction in mortality rates over the last decade, the mortality from heart failure continues to rise[1]. Thus, identifying novel therapies that can reduce heart failure development and/or progression are warranted. Unifying to most cardiomyopathic processes is an impaired handling of reactive oxygen species (ROS)[2-4]. Reactive oxygen species are generated as byproducts of inflammation and oxidative stress that occur in the setting of normal myocardial aerobic metabolism. Metallothionein, glutathione reductase, and superoxide dismutase are major antioxidants in the myocardium that help combat oxidative stress and prevent myocardial damage. In certain clinical settings, including cardiac ischemia, diabetes, and heavy metal excess (copper, iron), myocardial oxidative stress levels are greatly increased. When pro-oxidant levels exceed myocardial antioxidant capabilities, ROS-induced membrane, protein, and DNA inactivation can lead to the development of cardiac dysfunction.

One means of preventing the development or progression of cardiomyopathy is to reduce oxidative stress through up-regulation of intramyocardial antioxidants. Murine studies of cardiomyopathy have shown that oral administration of zinc acetate may succeed as an indirect myocardial anti-oxidant because zinc sufficiently up-regulates the intramyocardial production of superoxide dismutase (a zinc-dependant anti-oxidant enzyme) and metallothionein (a "super antioxidant") [5-8]. Zinc also directly reduces prooxidant Cu levels by reducing gastrointestinal zinc absorption. However, to date, no studies have examined the impact of zinc acetate supplementation in subjects with cardiomyopathy and systolic failure on antioxidant capacity and remodeling.

The hypothesis of this pilot study is that administration of oral zinc acetate to humans with cardiomyopathy will lead to an up-regulation of myocardial anti-oxidant capabilities,leading to a favorable reduction in oxidative stress. This study will provide preliminary data to support a randomized, placebo-controlled trial of zinc therapy in heart failure as a means of improving or preventing the progression of systolic dysfunction in subjects with mild-moderate heart failure.

DETAILED DESCRIPTION:
Altered regulation of the transition-metal copper (Cu) may lead to an overproduction of reactive oxygen species (ROS) with subsequent development of a nonischemic cardiomyopathy (NISCM). Myocardial Cu levels are elevated in NISCM, and Cu levels are highest in the "diabetic cardiomyopathy." In humans, zinc (Zn) is an essential component of proteins critical for regulating myocardial cytoskeleton turnover and cellular proliferation. Zn also serves as an antioxidant and indirect regulator of redox-active Cu. By upregulating the chelator metallothionein, Zn reduces the levels of free Cu implicated in oxidative myocardial damage.

Transgenic over-expression of the antioxidant metallothionein has been shown to reduce ROS-induced myocardial damage. In diabetic cardiomyopathy, Cu chelation improves left ventricular (LV) diastolic relaxation abnormalities. However, it is unknown if Zn supplementation could alter the progression of LV systolic dysfunction through Cu depletion and ROS reduction. The aim of this pilot study is to assess the impact of a novel intervention, Zn supplementation, on myocardial remodeling by examining changes in serum levels of the types I (PINP) and III (PIIINP) collagen N-terminal propeptides. The primary study hypothesis is that Zn supplementation will have a favorable impact on the pathophysiology of NISCM by either repleting a Zn deficiency/insufficiency or by reducing myocardial damage and adverse remodeling in the setting of redox-active Cu excess.

Stable outpatients (n=40) with chronic NISCM (ejection fraction ≤40%) will receive daily oral Zn-acetate (50 mg po tid) for 10 months. Serum PINP, PIIINP, and markers of inflammation (CRP, sedimentation rate, myeloperoxidase) and oxidative stress (8-isoprostane, superoxide dismutase) will be obtained at baseline and following 10 months of Zn supplementation. Changes in collagen turnover will then be correlated with changes noted in LV systolic and diastolic function by echocardiography. Finally, we will examine for a differential treatment effect of Zn therapy in a diabetic subset (n=20) with NISCM compared with the nondiabetics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (n=40) ≥21 years of age with chronic (≥1 year duration) nonischemic cardiomyopathy (NISCM), New York Heart Association (NYHA) functional class II-III symptoms on stable medical therapy (≥3 months of stable doses of β-blocker, angiotensin inhibitor or receptor blocker, and aldosterone inhibitor [if appropriate] therapies) with a documented left ventricular (LV) ejection fraction ≤40% and evidence of LV dilation will be eligible for study participation.
* The diagnosis of a nonischemic etiology for the cardiomyopathy must be supported by coronary angiography, stress echocardiography, or nuclear scintigraphy.
* To allow for a comparison of treatment effect in diabetic versus nondiabetic NISCM, half (n=20) of the subjects enrolled will be diabetic

Exclusion Criteria:

* Subjects with HF that is deemed to be ischemic, congenital, valvular, or infiltrative in etiology, or chemotherapy/toxin-induced will not be eligible for enrollment.
* Other exclusion criteria include the presence of a life-threatening illness with a projected survival ≤6 months;
* recurrent ventricular arrhythmias; end-stage renal failure;
* ongoing infection;
* inability to follow-up;
* collagen vascular disease (lupus, sarcoid);
* enrollment in another investigational study;
* unstable or symptomatic peripheral artery disease;
* prior or active Zn supplementation;
* or ongoing alcohol abuse.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Aaronson, MD, MS, Principal Investigator — University of Michigan; Jennifer A Cowger, MD, MS, Study Chair — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were mainly recruited from the University of Michigan outpatient Cardiovascular clinic. 10 healthy controls (to quantify "normal" values and QA laboratory results for novel measures) were recruited from the community via advertisement.
Pre-assignment Details: The study was intended to run for 6 months. After further discussion with experts in zinc therapy, we opted to extend the study to 10 months.
Groups:
- Zinc Acetate: The intervention group consisted of patients with heart failure. Patients were given Zinc Acetate 50 mg po three times a day for 10 months. The intended intervention group was n=40, of which n=38 were enrolled. Of these 38, n=25 completed 10 mo of follow-up.
- Control: The control group consistent of 10 persons without any known health conditions who provided laboratory samples at a single encounter to quantify "normal" values for the novel labs measured. No intervention was provided to the healthy controls.
Period: Overall Study
Arm/Group | Zinc Acetate | Control
Started | 38 | 10
Completed | 25 | 10
Not Completed | 13 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 8 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Controls: The control group consistent of 10 persons without any known health conditions who provided laboratory samples at a single encounter to quantify "normal" values for the novel labs measured. No intervention was provided to the healthy controls.
- Total: Total of all reporting groups
Arm/Group | Zinc Acetate | Controls | Total
Number analyzed (Participants) | 38 | 10 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (11) | 52 (8) | 55 (11)
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 64 years | 29 | 10 | 39
  >=65 years | 9 | 0 | 9
Sex/Gender, Customized [Number; unit: participants]
  Female | 10 | 6 | 16
  Male | 18 | 4 | 22
Region of Enrollment [Number; unit: participants]
  United States | 38 | 10 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Markers of Cardiac Collagen Turnover (PINP) in Patients With Systolic Heart Failure and Compared With Healthy Controls.
Description: The intervention group (patients with systolic heart failure) was given Zinc Acetate 50 mg po three times daily for 10 months. The change from baseline in markers of cardiac collagen turnover (PINP) in patients with systolic heart failure after 10 months of zinc acetate was measured and compared with a single measure from healthy controls.
Time Frame: Baseline (time 0) and after 10 months of Zinc Acetate.
Population: Power was determined using prior studies examining the change in PINP and (separately) PIIINP in heart failure following administration of aldactone. Results below are PINP. For Controls, a single measure was obtained without further followup.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- CHF Patients With Zinc Acetate: The intervention group (patients with systolic heart failure) was given Zinc Acetate 50 mg po three times a day for 10 months. The intended intervention group was n=40, of which n=38 were enrolled. Of these 38, n=25 completed 10 mo of follow-up.
- Healthy Controls: The control group consistent of 10 persons without any health conditions who provided laboratory samples to quantify "normal" values for the novel labs measured. No intervention was provided to the healthy controls. A single measure was obtained without further followup.
Arm/Group | CHF Patients With Zinc Acetate | Healthy Controls
Number analyzed (Participants) | 25 | 10
ng/ml
  PINP baseline (time 0): number analyzed (Participants) | 24 | 10
  PINP baseline (time 0) | 48.1 [41.6 to 68] | 48.1 [41.6 to 59.4]
  PINP after 10 mo therapy: number analyzed (Participants) | 25 | 0
  PINP after 10 mo therapy | 39 [31 to 53] |
Statistical Analysis 1: Comparison: CHF Patients With Zinc Acetate; p value represents test of paired (within patient) difference; Test type: Superiority or Other; p = 0.068, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: CHF Patients With Zinc Acetate vs Healthy Controls; p value tests difference between the marker in CHF patients at time 0 and Health Controls (between group); Test type: Superiority or Other; p = 0.022, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline in Serum Isoprostane in Patients With Systolic Heart Failure
Description: Change from baseline in serum isoprostane 10 months after Zn Acetate in patients with systolic heart failure and compared with a single measure in healthy subjects
Time Frame: Baseline (time 0) and 10 months
Population: power calculation using prior studies of the above laboratories. For Controls, a single measure was obtained without further followup.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- CHF Treated With Zinc Acetate: The intervention group (patients with systolic heart failure) was given Zinc Acetate 50 mg po three times a day for 10 months.
- Health Controls: The control group consistent of 10 persons without any health conditions who provided laboratory samples to quantify "normal" values for the novel labs measured. No intervention was provided to the healthy controls. A single measure was obtained without further followup.
Arm/Group | CHF Treated With Zinc Acetate | Health Controls
Number analyzed (Participants) | 25 | 10
pg/ml
  Isoprostane baseline: number analyzed (Participants) | 25 | 9
  Isoprostane baseline | 4.4 [3.4 to 5.3] | 3.8 [3.1 to 5.2]
  Isoprostane 10 mo: number analyzed (Participants) | 25 | 0
  Isoprostane 10 mo | 4.4 [3.3 to 5.3] |
Statistical Analysis 1: Comparison: CHF Treated With Zinc Acetate; p value represents test of paired (within patient) difference; Test type: Superiority or Other; p = 0.71, Sign test
Statistical Analysis 2: Comparison: CHF Treated With Zinc Acetate vs Health Controls; p value tests difference between the marker in CHF patients at time 0 and Health Controls (between group); Test type: Superiority or Other; p = 0.33, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: Change in PIIINP From Baseline After 10 Months of Zinc Acetate in Systolic Heart Failure and Compared With a Single Measure in Healthy Controls
Description: Change in PIIINP from baseline after 10 months of Zinc Acetate in patients with systolic heart failure and compared with a single measure in healthy controls
Time Frame: Baseline (time 0) and 10 months
Population: Specimens from healthy controls were only analyzed at one time frame.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- CHF Patients With Zinc Acetate: The intervention group (patients with systolic heart failure) was given Zinc Acetate 50 mg po three times a day for 10 months.
- Healthy Controls: The control group consistent of 10 persons without any health conditions who provided laboratory samples to quantify "normal" values for the novel labs measured. No intervention was provided to the healthy controls.
Arm/Group | CHF Patients With Zinc Acetate | Healthy Controls
Number analyzed (Participants) | 24 | 10
ng/ml
  PIIINP baseline | 5.3 [4.1 to 6.1] | 4.1 [3.1 to 4.5]
  PIIINP 10 months: number analyzed (Participants) | 24 | 0
  PIIINP 10 months | 5.3 [2.6 to 9] |
Statistical Analysis 1: Comparison: CHF Patients With Zinc Acetate; p value represents test of paired (within patient) difference; Test type: Superiority or Other; p = 0.69, Sign test
Statistical Analysis 2: Comparison: CHF Patients With Zinc Acetate vs Healthy Controls; p value tests difference between the marker in CHF patients at time 0 and Health Controls (between group); Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)

4. Other Pre Specified Outcome: Change From Baseline in Serum Superoxide Dismutase
Description: Change from baseline in serum superoxide dismutase after 10 months of zinc acetate in patients with systolic heart failure and compared with a single measure in healthy controls
Time Frame: Baseline (time 0) and 10 months
Population: Specimens from healthy controls were only analyzed at one time frame.
Measure: Median (Inter-Quartile Range); unit: units per microL
Groups:
- Health Controls: The control group consistent of 10 persons without any health conditions who provided laboratory samples to quantify "normal" values for the novel labs measured. No intervention was provided to the healthy controls.
Arm/Group | CHF Treated With Zinc Acetate | Health Controls
Number analyzed (Participants) | 25 | 10
units per microL
  SOD at Baseline | 160 [88 to 261] | 117 [40 to 262]
  SOD at 10 months: number analyzed (Participants) | 25 | 0
  SOD at 10 months | 151 [31 to 785] |
Statistical Analysis 1: Comparison: CHF Treated With Zinc Acetate; p value represents test of paired (within patient) difference; Test type: Superiority or Other; p = 0.48, Sign test
Statistical Analysis 2: Comparison: CHF Treated With Zinc Acetate vs Health Controls; p value tests difference between the marker in CHF patients at time 0 and Health Controls (between group); Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney)

5. Other Pre Specified Outcome: Change From Baseline in Serum Measures of of Myeloperoxidase (MPO) After 10 Months of Zinc Acetate Treatment
Description: Change from baseline in serum myeloperoxidase (MPO) after 10 months of zinc acetate treatment in patients with systolic heart failure and compared with a single measure from healthy controls
Time Frame: Baseline (time 0) and 10 months
Population: Healthy controls only analyzed at one time point
Measure: Median (Inter-Quartile Range); unit: units per L
Arm/Group | CHF Treated With Zinc Acetate | Health Controls
Number analyzed (Participants) | 24 | 10
units per L
  MPO baseline (time 0) | 455 [286 to 1212] | 295 [145 to 1061]
  MPO at 10 months: number analyzed (Participants) | 24 | 0
  MPO at 10 months | 816 [169 to 6294] |
Statistical Analysis 1: Comparison: CHF Treated With Zinc Acetate; p value represents test of paired (within patient) difference; Test type: Superiority or Other; p = 0.92, Sign test
Statistical Analysis 2: Comparison: CHF Treated With Zinc Acetate vs Health Controls; p value tests difference between the marker in CHF patients at time 0 and Health Controls (between group); Test type: Superiority or Other; p = 0.22, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event occurrences were captured at each follow-up visit and when notified by patients or patient's practitioner (if occurring outside of a standard follow-up visit).
Groups:
- HF Group: The zinc intervention group consisted of patients with heart failure who were provided zinc acetate for 10 months
- Healthy Controls: The control group consisted of 10 persons without any known health conditions who provided laboratory samples to quantify "normal" values for the novel labs measured. No intervention was provided to the healthy controls
Arm/Group | HF Group | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/38 | 0/10
Other Adverse Events (participants affected / at risk) | 6/38 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HF Group (N=38) | Healthy Controls (N=10)
Intracoronary stent (Cardiac disorders) | 1 (3) | 0 (0) — Deemed unlikely related to zinc therapy
Nonelective Hospitalization- accident (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) — bike accident with hospitalization
Nonelective Hospitalization- CHF exacerbation (Cardiac disorders) | 1 (3) | 0 (0) — Patient presented with abdominal pain and high BNP. Felt by outside hospital to have CHF exacerbation with RV CHF symptom predominance
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HF Group (N=38) | Healthy Controls (N=10)
dizziness (Nervous system disorders) | 1 (2) | 0 (0) — patient reported dizziness while taking zinc and voluntarily withdrew from the study
Odd taste in mouth (General disorders) | 1 (2) | 0 (0) — Patient did like the metallic taste in mouth and voluntarily withdrew from the study
Nausea (Gastrointestinal disorders) | 6 (6) | 0 (0) — 6 patients reported significant nausea taking the zinc acetate and 4 withdrew from the study due to nausea

LIMITATIONS AND CAVEATS:
Zinc acetate was poorly tolerated by some patients. Patients often commented on GI upset (nausea) and reflux symptoms at follow-up encounter. The myeloperoxidase assay demonstrated marked variability and test validity/quality is in question.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No